CLINICAL TRIAL: NCT02473536
Title: Safety Lead-in Phase II Trial of Neo-adjuvant SABR for IVC Tumor Thrombus in Newly Diagnosed RCC
Brief Title: Neo-adjuvant SABR for IVC Tumor Thrombus in Newly Diagnosed RCC
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Raquibul Hannan, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 022015-058
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: 6 for Lead-in phase; 23 for phase II
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic ablative radiation therapy (Experimental): SABR
  Interventions: Radiation: Stereotactic ablative radiation therapy

INTERVENTIONS:
Radiation: Stereotactic ablative radiation therapy — SABR

SUMMARY:
To evaluate the safety and feasibility of pre-operative SABR of RCC IVC tumor thrombus.

To evaluate the effect of pre-operative SABR in RCC IVC tumor thrombus on relapse free survival at one year.

DETAILED DESCRIPTION:
Stereotactic Ablative Radiation Therapy (SABR): 5 fractions of 8 Gy or 3 fractions of 12Gy. The concept of stereotactic radiosurgery involves tightly conforming dose of therapeutic radiation confined to a small region of the body. This results in eradication or ablation of the target tumor with sparing of surrounding normal tissues. The largest experience with stereotactic radiosurgery is for the treatment of intracranial tumors Neoadjuvant treatment of IVC-TT with SABR may decrease local recurrences and lower the likelihood of embolic complications and systemic metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Radiographic evidence of renal cancer with IVC tumor thrombus
2. Tumor thrombus must be ≥ level II (As per Mayo classification, it would be ≥ level I [Refer to NEVES, R. and ZINCKE, H. (1987), Surgical Treatment of Renal Cancer with Vena Cava Extension. British Journal of Urology, 59: 390-395. doi:10.1111/j.1464-410X.1987.tb04832.x])
3. Patient eligible for SABR to the IVC tumor thrombus as decided by the treating radiation oncologist
4. Patient eligible for IVC tumor thrombectomy as decided by the treating urologist
5. Any number of metastatic disease is allowed in the Pilot phase of the trial

   • For Phase II, metastatic patients will be allowed only if all sites of metastasis has been treated either surgically or radio-surgically (If limited sites of metastasis are present, all of which can be resected during the nephrectomy, then the patient can be eligible)
6. Age ≥ 18 years.
7. Performance status ECOG 0-2
8. Any serum Albumin is allowed, but ≥ 3.4 g/dL is strongly encouraged

   • Serum albumin <3.4 is a significant predictor of peri-operative mortality(12)
9. Any serum AST is allowed but serum AST ≤ 34 IU/L is strongly encouraged

   • Significant predictor of mortality in univariate but not multivariate analysis(12)
10. Women of childbearing potential and men must agree to use adequate contraception (hormonal such as birth control pills, patch or ring; Depo-Provera, Implanon or barrier method, such as condom or diaphragm used with a spermicide of birth control; abstinence) prior to study entry, for the duration of study treatment, and for 90 days following completion of radiation therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

    10.1 A female of childbearing potential is any woman (regardless of sexual orientation, marital status, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
    * Has not undergone a hysterectomy or bilateral oophorectomy; or
    * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
11. Ability to understand and the willingness to sign a written informed consent.
12. Subjects must be able to undergo either MRI or CT.

Exclusion Criteria:

1. Subjects who have had radiotherapy to a target within 3 cm of the IVC tumor thrombus.
2. Subjects may have received any other investigational agents or chemotherapy as long as they are eligible for SABR and surgery
3. Subjects with brain metastases should be excluded from this clinical trial unless all the metastasis are treated surgically or radio-surgically
4. Subjects with a history of pulmonary embolism is excluded
5. Subjects with a history of pulmonary hypertension is excluded
6. Subjects must not be pregnant due to the potential for congenital abnormalities.
7. Contraindication for contrast-enhanced MRI as defined by the standard operating procedures of the Department of Radiology at UT Southwestern. Briefly, these include medically unstable; cardiac pacemaker; intracranial clips, metal implants; metal in the eyes; pregnant or nursing; claustrophobia; and impairment of the renal function with estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2. Patients with one or more of these contraindications but eligible to undergo contrast-enhanced CT can participate in this study and will not receive an MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
To determine the feasibility of neoadjuvant SABR followed immediately by IVC tumor thrombectomy | 90 days
  The treatment duration will be between 2-3 weeks depending on the fraction scheme chosen.
To determine the operative safety of neoadjuvant SABR followed immediately by IVC tumor thrombectomy | 90 days
  The treatment duration will be between 2-3 weeks depending on the fraction scheme chosen.
Survival at one year | ONE YEAR
  Phase II To determine the relapse-free survival at one-year

SECONDARY OUTCOMES:
Peri-operative morbidity | 90 days
  To describe the associated peri-operative morbidity. Associated peri-operative morbidity is defined as grade>2 side effects as assessed by NCI's CTCAE v4.0 toxicity within one year of surgery.
Adverse events post surgery | 1 year
  To determine the associated adverse events within one year of surgery. Associated adverse events are any toxicity as defined by NCI's CTCAE v4.0 toxicity criteria for the first year post- surgery.
Recurrence free survival (1 year) | 1 year
  To determine the 1 year recurrence free survival
Recurrence free survival overall | 7 years
  To determine the recurrence free survival
Recurrence | 7 years
  To determine the median time to recurrence
Pulmonary emboli | 1 year
  To determine the rate of pulmonary emboli within one year of surgery. Pulmonary Emboli: Pulmonary embolus determined in patients that become symptomatic and as a result has radiographic evidence of pulmonary embolus on CT angio or V/Q scan.
Pulmonary metastasis | 7 years
  To determine the rate of pulmonary metastasis. Pulmonary Metastasis: Any evidence of new lung metastasis >1.0 cm
  • New lung nodules >0.5cm will also be reported.
Systemic metastasis | 7 years
  To determine the rate of systemic metastasis. Systemic Metastasis: Any evidence of new metastasis that is progressing on a second scan > 6 weeks apart
Overall survival | 7 years
  The rate of overall survival. Overall Survival: Time to death from the date of treatment start.

CONTACTS AND LOCATIONS:
Overall Officials: Raquibul Hannan, MD, Principal Investigator — UTSW
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No